CLINICAL TRIAL: NCT04318366
Title: Study to Characterize Patients With SARS-Cov-2 Infection and to Create a Biobank to Identify Predictors of Disease Severity, Mortality and Treatment Response
Brief Title: COVID-19 Patients Characterization, Biobank, Treatment Response and Outcome Predictor
Acronym: COVID-BioB
Status: Recruiting | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Associate Professor, Università Vita-Salute San Raffaele
Other Study IDs: COVID-BioB/OSR
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Coronavirus Infections
MeSH Terms: conditions — Coronavirus Infections | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study — Not required

SUMMARY:
Collection and analysis of demographic, clinical, radiographic and laboratory characteristics of CoViD-19 patients to identify predictors of disease severity, mortality and treatment response, and to identify subgroup of patients that might benefit from specific therapeutic interventions

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to hospital with biological samples positive for SARS-CoV-2
* Patients admitted to hospital with negative test but clinical and radiological characteristics highly suggestive of SARS-CoV-2 disease
* Patients discharged from emergency department with biological samples positive for SARS-CoV-2

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-03-19 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Characterize Patients With SARS-Cov-2 Infection and to Create a Biobank to Identify Predictors of Disease Severity, Mortality and Treatment Response | Hospital stay (2-3 weeks)
  Characterize Patients With SARS-Cov-2 Infection and to Create a Biobank to Identify Predictors of Disease Severity, Mortality and Treatment Response

CONTACTS AND LOCATIONS:
Locations (13):
- Italy (13):
  - Autoimmunity and Vascular Inflammation Unit, Division of Regenerative Medicine, Stem Cells and Gene Therapy - IRCCS San Raffaele Scientific Institute, Milan, Lombardy
  - AIDS Immunopathogenesis Unit - IRCCS San Raffaele Scientific Institute, Milan, Lombardy
  - Department of Infection Diseases - IRCCS San Raffaele Scientific Institute -, Milan, Lombardy
  - Department of Internal Medicine - IRCCS San Raffaele Scientific Institute, Milan, Lombardy
  - Diabetes Research Institute -IRCCS San Raffaele Scientific Istitute, Milan, Lombardy
  - Division of Immunology, Transplantation and Infectious Diseases - IRCCS San Raffaele Scientific Institute, Milan, Lombardy
  - Division of Research of Regenerative Medicine, Cell and Gene Therapy - IRCCS San Raffaele Scientific Istitute, Milan, Lombardy
  - Laboratory of Microbiology and Virology - IRCCS San Raffaele Scientific Institute, Milan, Lombardy
  - Nephrology Unit - IRCCS San Raffaele Scientific Institute, Milan, Lombardy
  - Strategic Program in Nephrology and Dialysis - IRCCS San Raffaele Scientific Institute, Milan, Lombardy
  - Viral pathogens and biosafety Unit - IRCCS San Raffaele Scietific Institute, Milan, Lombardy
  - Unit of Immunology, Rheumatology, Allergy and Rare Diseases - IRCCS San Raffaele Scientific Institute, Milan, Lombardy
  - Università Vita-Salute San Raffaele, Milan, Mi

REFERENCES:
- [Background] Ciceri F, Beretta L, Scandroglio AM, Colombo S, Landoni G, Ruggeri A, Peccatori J, D'Angelo A, De Cobelli F, Rovere-Querini P, Tresoldi M, Dagna L, Zangrillo A. Microvascular COVID-19 lung vessels obstructive thromboinflammatory syndrome (MicroCLOTS): an atypical acute respiratory distress syndrome working hypothesis. Crit Care Resusc. 2020 Apr 15;22(2):95-97. doi: 10.51893/2020.2.pov2. Online ahead of print. PMID 32294809
- [Derived] Merolla A, De Lorenzo R, Paolazzi G, Critelli S, Palladini M, Damanti S, Vitali G, Canti V, Cilla M, Martinenghi S, Falbo E, Ferrante M, Castellani J, Pacioni G, Magnaghi C, Fumagalli A, Mazza MG, Benedetti F, Rovere-Querini P. Micronized/ultramicronized palmitoylethanolamide improves depression and fatigue in coronavirus disease 2019 (COVID-19) survivors. Int Clin Psychopharmacol. 2024 Nov 1;39(6):361-368. doi: 10.1097/YIC.0000000000000537. Epub 2024 Feb 22. PMID 38381905
- [Derived] Zangrillo A, Colombo S, Scandroglio AM, Fominskiy E, Pieri M, Calabro MG, Beccaria PF, Pasculli N, Guzzo F, Calvi MR, Cipriani A, Sartini C, Nardelli P, Ortalda A, Lombardi G, Sartorelli M, Monti G, Assanelli A, Tresoldi M, Dagna L, Franchini S, Neto AS, Bellomo R, Landoni G. Angiotensin II infusion and markers of organ function in invasively ventilated COVID-19 patients. Crit Care Resusc. 2023 Oct 18;23(2):215-224. doi: 10.51893/2021.2.oa9. eCollection 2021 Jun. PMID 38045523
- [Derived] Negro A, Villa G, Cardinali M, Gianelle N, Ranzani R, Rolandi S, Maimeri N, Zangrillo A. Is Gastrointestinal Bleeding a Problem for COVID-19 Intensive Care Unit Patients? Gastroenterol Nurs. 2023 May-Jun 01;46(3):225-231. doi: 10.1097/SGA.0000000000000722. Epub 2023 Apr 11. PMID 37053376
- [Derived] De Lorenzo R, Palmisano A, Esposito A, Gnasso C, Nicoletti V, Leone R, Vignale D, Falbo E, Ferrante M, Cilla M, Magnaghi C, Martinenghi S, Vitali G, Molfino A, Rovere-Querini P, Muscaritoli M, Conte C. Myosteatosis Significantly Predicts Persistent Dyspnea and Mobility Problems in COVID-19 Survivors. Front Nutr. 2022 Apr 8;9:846901. doi: 10.3389/fnut.2022.846901. eCollection 2022. PMID 35464004
- [Derived] Dispinseri S, Marzinotto I, Brigatti C, Pirillo MF, Tolazzi M, Bazzigaluppi E, Canitano A, Borghi M, Gallinaro A, Caccia R, Vercesi R, McKay PF, Ciceri F, Piemonti L, Negri D, Cinque P, Cara A, Scarlatti G, Lampasona V. Seasonal Betacoronavirus Antibodies' Expansion Post-BNT161b2 Vaccination Associates with Reduced SARS-CoV-2 VoC Neutralization. J Clin Immunol. 2022 Apr;42(3):448-458. doi: 10.1007/s10875-021-01190-5. Epub 2022 Jan 9. PMID 35000058
- [Derived] Conte C, Esposito A, De Lorenzo R, Di Filippo L, Palmisano A, Vignale D, Leone R, Nicoletti V, Ruggeri A, Gallone G, Secchi A, Bosi E, Tresoldi M, Castagna A, Landoni G, Zangrillo A, De Cobelli F, Ciceri F, Camici P, Rovere-Querini P. Epicardial adipose tissue characteristics, obesity and clinical outcomes in COVID-19: A post-hoc analysis of a prospective cohort study. Nutr Metab Cardiovasc Dis. 2021 Jun 30;31(7):2156-2164. doi: 10.1016/j.numecd.2021.04.020. Epub 2021 May 3. PMID 34059384
- [Derived] Di Filippo L, De Lorenzo R, Cinel E, Falbo E, Ferrante M, Cilla M, Martinenghi S, Vitali G, Bosi E, Giustina A, Rovere-Querini P, Conte C. Weight trajectories and abdominal adiposity in COVID-19 survivors with overweight/obesity. Int J Obes (Lond). 2021 Sep;45(9):1986-1994. doi: 10.1038/s41366-021-00861-y. Epub 2021 May 17. PMID 34002039
- [Derived] Vanella G, Capurso G, Burti C, Fanti L, Ricciardiello L, Souza Lino A, Boskoski I, Bronswijk M, Tyberg A, Krishna Kumar Nair G, Angeletti S, Mauro A, Zingone F, Oppong KW, de la Iglesia-Garcia D, Pouillon L, Papanikolaou IS, Fracasso P, Ciceri F, Rovere-Querini P, Tomba C, Viale E, Eusebi LH, Riccioni ME, van der Merwe S, Shahid H, Sarkar A, Yoo JWG, Dilaghi E, Speight RA, Azzolini F, Buttitta F, Porcari S, Petrone MC, Iglesias-Garcia J, Savarino EV, Di Sabatino A, Di Giulio E, Farrell JJ, Kahaleh M, Roelandt P, Costamagna G, Artifon ELA, Bazzoli F, Testoni PA, Greco S, Arcidiacono PG. Gastrointestinal mucosal damage in patients with COVID-19 undergoing endoscopy: an international multicentre study. BMJ Open Gastroenterol. 2021 Feb;8(1):e000578. doi: 10.1136/bmjgast-2020-000578. PMID 33627313
- [Derived] Di Filippo L, De Lorenzo R, D'Amico M, Sofia V, Roveri L, Mele R, Saibene A, Rovere-Querini P, Conte C. COVID-19 is associated with clinically significant weight loss and risk of malnutrition, independent of hospitalisation: A post-hoc analysis of a prospective cohort study. Clin Nutr. 2021 Apr;40(4):2420-2426. doi: 10.1016/j.clnu.2020.10.043. Epub 2020 Oct 29. PMID 33160700
- [Derived] Secchi M, Bazzigaluppi E, Brigatti C, Marzinotto I, Tresoldi C, Rovere-Querini P, Poli A, Castagna A, Scarlatti G, Zangrillo A, Ciceri F, Piemonti L, Lampasona V. COVID-19 survival associates with the immunoglobulin response to the SARS-CoV-2 spike receptor binding domain. J Clin Invest. 2020 Dec 1;130(12):6366-6378. doi: 10.1172/JCI142804. PMID 32991329
- [Derived] Mushtaq J, Pennella R, Lavalle S, Colarieti A, Steidler S, Martinenghi CMA, Palumbo D, Esposito A, Rovere-Querini P, Tresoldi M, Landoni G, Ciceri F, Zangrillo A, De Cobelli F. Initial chest radiographs and artificial intelligence (AI) predict clinical outcomes in COVID-19 patients: analysis of 697 Italian patients. Eur Radiol. 2021 Mar;31(3):1770-1779. doi: 10.1007/s00330-020-07269-8. Epub 2020 Sep 18. PMID 32945968
- [Derived] Zangrillo A, Beretta L, Scandroglio AM, Monti G, Fominskiy E, Colombo S, Morselli F, Belletti A, Silvani P, Crivellari M, Monaco F, Azzolini ML, Reineke R, Nardelli P, Sartorelli M, Votta CD, Ruggeri A, Ciceri F, De Cobelli F, Tresoldi M, Dagna L, Rovere-Querini P, Serpa Neto A, Bellomo R, Landoni G; COVID-BioB Study Group. Characteristics, treatment, outcomes and cause of death of invasively ventilated patients with COVID-19 ARDS in Milan, Italy. Crit Care Resusc. 2020 Sep;22(3):200-211. doi: 10.1016/S1441-2772(23)00387-3. PMID 32900326
- [Derived] Pagnesi M, Baldetti L, Beneduce A, Calvo F, Gramegna M, Pazzanese V, Ingallina G, Napolano A, Finazzi R, Ruggeri A, Ajello S, Melisurgo G, Camici PG, Scarpellini P, Tresoldi M, Landoni G, Ciceri F, Scandroglio AM, Agricola E, Cappelletti AM. Pulmonary hypertension and right ventricular involvement in hospitalised patients with COVID-19. Heart. 2020 Sep;106(17):1324-1331. doi: 10.1136/heartjnl-2020-317355. Epub 2020 Jul 16. PMID 32675217
- [Derived] Cavalli G, De Luca G, Campochiaro C, Della-Torre E, Ripa M, Canetti D, Oltolini C, Castiglioni B, Tassan Din C, Boffini N, Tomelleri A, Farina N, Ruggeri A, Rovere-Querini P, Di Lucca G, Martinenghi S, Scotti R, Tresoldi M, Ciceri F, Landoni G, Zangrillo A, Scarpellini P, Dagna L. Interleukin-1 blockade with high-dose anakinra in patients with COVID-19, acute respiratory distress syndrome, and hyperinflammation: a retrospective cohort study. Lancet Rheumatol. 2020 Jun;2(6):e325-e331. doi: 10.1016/S2665-9913(20)30127-2. Epub 2020 May 7. PMID 32501454